CLINICAL TRIAL: NCT02620852
Title: Enabling a Paradigm Shift: A Preference-Tolerant RCT of Personalized vs. Annual Screening for Breast Cancer (Wisdom Study)
Brief Title: Women Informed to Screen Depending on Measures of Risk (Wisdom Study)
Acronym: WISDOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Robert Wood Johnson Foundation (Other); Color Genomics, Inc. (Industry); Salesforce (Unknown); National Cancer Institute (NCI) (NIH); Safeway Foundation (Unknown); United States Department of Defense (U.S. Federal Agency); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PCS-1402-10749; NCI-2018-00562 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R01CA237533-01A1 (NIH); 16752 (Other: University of California, San Francisco)
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Screening; Breast Carcinoma in Situ; Breast Cancer
Keywords: Breast screening; mammography; prevention; risk assessment; DCIS; Breast cancer; Wisdom
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Annual Arm (Active Comparator): Women in this arm will receive Athena standard of care mammography screening, including annual mammograms. They will complete a health questionnaire and receive screening advice based on a basic risk assessment.
  Interventions: Other: Complete a health questionnaire; Other: Screening advice based on a basic risk assessment
- Risk-Based Arm (Experimental): Women in this arm will receive risk-based screening, where risk is calculated based on a model including personal history, family history, and genetic testing. All women in the risk-based arm complete a health questionnaire, provide a saliva sample for genetic testing, and receive screening advice based on a comprehensive risk assessment. Women in this arm will be tested for a panel of 9 genes related to breast cancer risk as well as a panel of SNPs, which can further modify risk. Women will be assigned a screening start date, screening stop date, and screening frequency.
  Interventions: Other: Complete a health questionnaire; Device: Provide a saliva sample for genetic testing; Other: Screening advice based on a comprehensive risk assessment

INTERVENTIONS:
Other: Complete a health questionnaire — Complete a health history questionnaire.
Device: Provide a saliva sample for genetic testing — Provide a saliva sample for testing of 9 genes and a panel of single nucleotide polymorphisms (SNPs) that influence breast cancer risk
  Arms: Risk-Based Arm
Other: Screening advice based on a comprehensive risk assessment — Receive a screening schedule recommendation
  Arms: Risk-Based Arm
Other: Screening advice based on a basic risk assessment — Receive a screening schedule recommendation
  Arms: Annual Arm

SUMMARY:
Most physicians still use a one-size-fits-all approach to breast screening in which all women, regardless of their personal history, family history or genetics (except BRCA carriers) are recommended to have annual mammograms starting at age 40. Mammograms benefit women by detecting cancers early when they are easier to treat, but they are not perfect. Recent news stories have discussed some of the potential harms: large numbers of positive results that cause stressful recalls for additional mammograms and biopsies. With the current screening approach, half of the women who undergo annual screening for ten years will have at least one false positive biopsy. Potentially more important are cancer diagnoses for growths that might never come to clinical attention if left alone (called "overdiagnosis"). This can lead to unnecessary treatment. Even more concerning is evidence that up to 20% of breast cancers detected today may fall into the category of "overdiagnosis."

The WISDOM 1.0 study compares annual screening with a risk-based breast cancer screening schedule, based upon each woman's personal risk of breast cancer. The investigators have designed the study to be inclusive of all, so that even women who might be nervous about being randomly assigned to receive a particular type of care (a procedure that is typical in clinical studies) will still be able to participate by choosing the type of care they receive.

For participants in the risk-based screening arm, each woman will receive a personal risk assessment that includes her family and medical history, breast density measurement and tests for genes (mutations and variations) linked to the development of breast cancer. Women who have the highest personal risk of developing breast cancer will receive more frequent screening, while women with a lower personal risk would receive less frequent screening. No woman will be screened less than is recommended by the USPSTF breast cancer screening guidelines.

If this study is successful, women will gain a realistic understanding of their personal risk of breast cancer as well as strategies to reduce their risk, and fewer women will suffer from the anxiety of false positive mammograms and unnecessary biopsies. The investigators believe this study has the potential to transform breast cancer screening in America.

Starting in Spring 2023, WISDOM's design shifted to remove the randomized option, but will continue with the preference/self-selection option for participation (WISDOM 2.0). Participants will therefore continue to choose their study arm (Personalized or Annual) rather than have the option to be randomized. This study design change was made after review of the WISDOM 1.0 data by an independent monitoring committee, which indicates that personalized screening does not cause harm. WISDOM 2.0 has also lowered the eligibility to ages 30-74. Women ages 30-39 will only be offered to join the Personalized Arm.

DETAILED DESCRIPTION:
For almost 30 years, annual mammograms for women over 40 have been a cornerstone of the US strategy to reduce mortality from breast cancer. A number of advances in the understanding of breast cancer biology, and screening in general, have led to calls to revise and improve national screening strategies (Esserman et al., 2014). In 2009, the US Preventive Services Task Force (USPSTF) introduced changes to screening guidelines, recommending that annual mammograms for all women 40-75 be replaced by biennial screening for women ages 50-75, and that screening in the 40's should be individualized by taking patient context into account, including the patient's values regarding specific benefits and harms. Despite being based on a thorough review of the scientific literature, these recommendations continue to spark debate and scientific opinion on the effectiveness of annual screening is greatly divided. On one hand the radiology and obstetrics/gynecology community argues that annual mammograms starting at 40 reduce the rate of interval cancers. On the other hand, primary care physicians and other specialists believe that annual screening results in more false-positives and unnecessary treatment and that a more targeted approach could result in fewer false-positives and less over-diagnosis without increasing the number of interval cancers. In fact it has been estimated that half of women will receive a false-positive recall over 10 years of annual screening and that as many as 20% of all breast cancers might be overdiagnosed. Since 2009 this debate has intensified, paralyzing the system and thwarting any efforts to change or improve screening. The end result is that women are frustrated and confused, and some have stopped screening altogether.

Despite a vastly improved understanding of breast cancer risk, the only criteria used to establish a woman's screening recommendations is her age (and BRCA status if known), but there are risk models available that incorporate personal and family history of breast disease, endocrine exposures and breast density to assess breast cancer risk (Constantino, et al., 1999; Parmigiani, et al., 1998; Tyrer, et al., 2004; Claus, et al., 2001; Ozanne, et al., 2003). Most recently certain genetic mutations and common genetic variants (single nucleotide polymorphisms or SNPs) have been confirmed predictors as well (Darabi, et al., 2012). Therefore, advances in this understanding of breast cancer biology, risk assessment, and imaging have enabled the creation of better tools and sufficient knowledge to replace the one-size-fits-all approach to screening and to implement a new, personalized model; one that provides recommendations on when to start, when to stop, and how often to screen that depend upon well characterized measures of risk.

The investigators propose to test a transformational evidence-based approach to breast screening that educates women about their actual risk, and tailors screening recommendations to them as individuals. Within the Athena Breast Health Network, the study will compare comprehensive, patient-centered risk-based screening to annual screening for women starting at age 40. The comprehensive risk assessment is based on a widely accepted risk model, the Breast Cancer Surveillance Consortium model, that includes endocrine exposures, family history and breast density, with additional genomic risk factors that include rare and uncommon major breast cancer susceptibility alleles as well as more common and recently validated single nucleotide polymorphisms (SNPs) that can, cumulatively, contribute significantly to a woman's individual risk. The study's personalized approach will recommend an age to start and stop screening as well as a frequency based upon individual risk. Women of highest risk will receive greater surveillance than those of lowest risk where the lower bound is the USPSTF recommended guidelines. In this manner, the study will focus the most effort on those most likely to develop the disease.

In close collaboration with patient advocates, the WISDOM 1.0 study has been designed as a 5-year, preference-tolerant, 65,000 patient, randomized controlled trial of risk-based versus annual screening. Individuals uncomfortable with the potential to be assigned to a particular arm in the randomized cohort can participate in the self-assigned observational cohort, an example of the pragmatic approach taken. Total accrual is anticipated to be 100,000 women across both cohorts. A broad group of stakeholders have participated in crafting this approach, including advocates, payers, the entire range of medical specialists and primary care providers and researchers involved with breast cancer screening across the entire Athena Network, technology partners, the Office of the President at the University of California, and policy-making organizations. WISDOM 1.0 trial was originally designed to randomize 65,000 women and be completed after five years to provide a median of ~3 years of exposure time in each randomized arm. However, due to slow initial accrual, trial duration was extended to up to ten years enabling a sample size reduction with maintained statistical power. The accrual goals were updated and approved by the DSMB and the Patient Centered Outcomes Research Institute.

The study hypothesizes that risk-based screening will be an improvement over annual screening because it will be as safe, less morbid, enable more cancer prevention, less stressful and more readily accepted by women as a result of an improved understanding of their personal risk.

The Athena Breast Health Network was established across the 5 University of California medical centers to develop a new, harmonized approach to breast cancer prevention, screening and treatment. Athena is among the few centers in North America to use technology to integrate risk assessment into breast screening. The investigators have developed a cadre of "breast health specialists" who provide women with counseling and support around risk and prevention. There are currently 100,000 registered Athena participants, with 30,000 new patients per year and growing with the addition of Sanford Health, one of the largest rural health networks in the country. The primary research mission of Athena is to address issues requiring a population-based approach and translate solutions to clinical practice. Athena is uniquely positioned to address the screening controversy and provide women with renewed confidence in decisions about their breast health. Risk-based screening for breast cancer is exactly the advanced, evidence-based approach to medicine described in the NIH and FDA's "Path to Personalized Medicine". If these hypotheses prove to be correct, this study will be able to establish a clear justification for its use, and provide a framework for widespread implementation that will benefit women across the country.

Starting in Spring 2023, WISDOM's design shifted to remove the randomized option, but will continue with the preference/self-selection option for participation (WISDOM 2.0). Participants will therefore continue to choose their study arm (Personalized or Annual) rather than have the option to be randomized. This study design change was made after review of the WISDOM 1.0 data by an independent monitoring committee, which indicates that personalized screening does not cause harm. WISDOM 2.0 has also lowered the eligibility to ages 30-74. Women ages 30-39 will only be offered to join the Personalized Arm.

ELIGIBILITY:
Inclusion Criteria:

1. Female*
2. Age 30 years to 74 years old**
3. Reside in the United States***

NOTE*: As of 2019, we are now enrolling all persons who identify as female, and will capture both their sex at birth and gender identity in the baseline survey.

NOTE**: Eligibility from 2016 - October 2023 included ages 40-74 (WISDOM 1.0) and expanded to age 30 in October 2023 (WISDOM 2.0).

NOTE***: As of 2019, recruitment is available nationwide. Original eligibility was limited to California, North Dakota, South Dakota, Iowa, Minnesota, Alabama, Louisiana, Illinois OR have coverage from a participating health plan.

Exclusion Criteria:

1. Prior Breast cancer or ductal carcinoma in situ (DCIS) diagnosis
2. Prior prophylactic bilateral mastectomy
3. Inability to provide consent
4. Non-English or Spanish proficiency (Spanish participation available: June 2019)

Ages: 30 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2016-08-31 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Late-stage cancer | 5 years (minimum)
  Proportion of cancers diagnosed at Stage IIB or higher
Biopsy rate | 5 years (minimum)
  Rate of biopsies performed

SECONDARY OUTCOMES:
Late-stage cancer rate and interval cancer rate | 5 years (minimum)
  Rate of Stage IIB or higher cancers and rate of interval (detected within 12-24 months of a normal screen) cancers
Rate of stage IIA cancers | 5 years (minimum)
  To assess the difference between the arms in the rate of stage IIA cancers (prognostic and anatomic), specifically to test for non-inferiority of personalized screening compared with annual screening with respect to detection rates of prognostic and anatomic stage IIA cancers.
Rate of systemic therapy | 5 years (minimum)
  Rate of systemic therapy as measure of morbidity
Breast imaging rate | 5 years (minimum)
  Breast imaging (Mammogram or MRI) rate as measure of morbidity
Breast biopsy rate | 5 years (minimum)
  Breast biopsy rate as measure of morbidity
DCIS rate | 5 years (minimum)
  Rate of ductal carcinoma in situ (DCIS) as a measure of morbidity, stratified by biologic type
Chemoprevention uptake rate | 5 years (minimum)
  Rate of uptake of endocrine prevention interventions
Choice of risk-based versus annual screening in self-assigned cohort | 5 years (minimum)
  Proportion of participants who choose risk-based versus annual screening in the self-assigned cohort as a measure of acceptability
Adherence to assigned screening schedule | 5 years (minimum)
  Proportion of participants who adhere to their assigned screening schedules as a measure of acceptability
Breast-cancer anxiety | 5 years (minimum)
  Breast cancer anxiety (as measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety scale) as a measure of acceptability
Decisional regret | 5 years (minimum)
  Decisional regret (as measured with the Decision Regret Scale, a 5-item Likert scale) as a measure of acceptability
Ultra-low risk cancer rate | 5 years (minimum)
  Rates of ultra-low risk cancer

CONTACTS AND LOCATIONS:
Overall Officials: Laura Esserman, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Irvine, Irvine, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - TopLine MD Alliance, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Louisiana State University, New Orleans, Louisiana
  - Weill Cornell Medicine, New York, New York
  - Edith Sanford Breast Center, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esserman LJ, Thompson IM, Reid B, Nelson P, Ransohoff DF, Welch HG, Hwang S, Berry DA, Kinzler KW, Black WC, Bissell M, Parnes H, Srivastava S. Addressing overdiagnosis and overtreatment in cancer: a prescription for change. Lancet Oncol. 2014 May;15(6):e234-42. doi: 10.1016/S1470-2045(13)70598-9. PMID 24807866
- [Background] Costantino JP, Gail MH, Pee D, Anderson S, Redmond CK, Benichou J, Wieand HS. Validation studies for models projecting the risk of invasive and total breast cancer incidence. J Natl Cancer Inst. 1999 Sep 15;91(18):1541-8. doi: 10.1093/jnci/91.18.1541. PMID 10491430
- [Background] Parmigiani G, Berry D, Aguilar O. Determining carrier probabilities for breast cancer-susceptibility genes BRCA1 and BRCA2. Am J Hum Genet. 1998 Jan;62(1):145-58. doi: 10.1086/301670. PMID 9443863
- [Background] Tyrer J, Duffy SW, Cuzick J. A breast cancer prediction model incorporating familial and personal risk factors. Stat Med. 2004 Apr 15;23(7):1111-30. doi: 10.1002/sim.1668. PMID 15057881
- [Background] Claus EB. Risk models used to counsel women for breast and ovarian cancer: a guide for clinicians. Fam Cancer. 2001;1(3-4):197-206. doi: 10.1023/a:1021135807900. PMID 14574179
- [Background] Ozanne EM, Annis C, Adduci K, Showstack J, Esserman L. Pilot trial of a computerized decision aid for breast cancer prevention. Breast J. 2007 Mar-Apr;13(2):147-54. doi: 10.1111/j.1524-4741.2007.00395.x. PMID 17319855
- [Background] Darabi H, Czene K, Zhao W, Liu J, Hall P, Humphreys K. Breast cancer risk prediction and individualised screening based on common genetic variation and breast density measurement. Breast Cancer Res. 2012 Feb 7;14(1):R25. doi: 10.1186/bcr3110. PMID 22314178
- [Derived] Fergus KB, Ross KS, Scheuner MT, Blanco AM, Tice JA, Ziv E, Shieh Y, van 't Veer L, Olopade OI, Goodman DL, Tong BS, Harvey H, DeRosa D, Risty L, Silver E, Kaster A, Fiscalini AS, Blum K, Heise R, Sabacan L, Heditsian D, Brain S, Petruse A, Eklund M, Hiatt RA, Borowsky AD, Naeim A, Park HL, LaCroix AZ, Parker BA, Lancaster R, Esserman J, Wenger N, Arasu V, Anton-Culver H, Esserman LJ, Madlensky L. Germline Pathogenic Variants Among Women Without a History of Breast Cancer: A Secondary Analysis of the WISDOM Randomized Clinical Trial. JAMA Intern Med. 2025 Dec 12:e257323. doi: 10.1001/jamainternmed.2025.7323. Online ahead of print. PMID 41385723
- [Derived] Esserman LJ, Fiscalini AS, Naeim A, Van't Veer LJ, Kaster A, Scheuner MT, LaCroix AZ, Borowsky AD, Anton-Culver H, Olopade OI, Esserman J, Lancaster R, Madlensky L, Blanco AM, Ross KS, Goodman DL, Tong BS, Hogarth M, Heditsian D, Brain S, Lee V, Blum K, Kim MO, Sabacan LP, Fergus KB, Yau C, Park HL, Parker BA, Kaplan C, Rhoads KF, Eder S, Adduci K, Matthews JB, Wenger NS, Shieh Y, Hiatt RA, Ziv E, Tice JA, Eklund M. Risk-Based vs Annual Breast Cancer Screening: The WISDOM Randomized Clinical Trial. JAMA. 2025 Dec 12:e2524784. doi: 10.1001/jama.2025.24784. Online ahead of print. PMID 41385349
- [Derived] Fergus KB, Heise RS, Madlensky L, Fiscalini A, Sabacan L, Theiner S, Kapoor S, Soto IA, Blanco A, Ross K, Goodman-Gruen D, Scheuner M, Hu D, Heditsian D, Brain S, Arasu VA, Kaster A, Chapa L, Olopade OI, Eklund M, Tice JA, Ziv E, van 't Veer L, Esserman LJ, Shieh Y; Athena/WISDOM Network Collaborators and Advocate Partners. Integrating breast cancer polygenic risk scores at scale in the WISDOM Study: a national randomized personalized screening trial. Genome Med. 2025 Aug 28;17(1):97. doi: 10.1186/s13073-025-01524-7. PMID 40877879
- [Derived] Leggat-Barr K, Ryu R, Hogarth M, Stover-Fiscalini A, Veer LV', Park HL, Lewis T, Thompson C, Borowsky A, Hiatt RA, LaCroix A, Parker B, Madlensky L, Naeim A, Esserman L. Early Ascertainment of Breast Cancer Diagnoses Comparing Self-Reported Questionnaires and Electronic Health Record Data Warehouse: The WISDOM Study. JCO Clin Cancer Inform. 2023 Aug;7:e2300019. doi: 10.1200/CCI.23.00019. PMID 37607323